CLINICAL TRIAL: NCT03758976
Title: SCAN-B-rec: Infrastructure, Technology Platform and Clinical Research Development to Profile and Monitor Metastatic Breast Cancer
Brief Title: Sweden Cancerome Analysis Network - Breast Recurrence (SCAN-B-rec)
Status: Recruiting | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCAN-B-rec
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Molecular profiling; Circulating tumor DNA; Circulating tumor cells
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tissue biopsy, whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biopsies, blood — We will perform targeted exon sequencing on paraffin embedded tissues from metastatic breast cancer
  Other Names: Targeted exon sequencing

SUMMARY:
Prospective multicenter observational study to assess molecular drivers of metastatic breast cancer and disease evolution upon therapeutic pressure.

The main aim is to develop and validate prognostic, predictive and pathogenic markers in clinically well-characterized population-based material of breast cancer tumors and the corresponding normal tissue.These data will be used to characterize recurrent breast cancer on a molecular level, study tumor evolution, develop biomarkers of response/resistance to targeted therapy in the metastatic setting, enroll patients on targeted treatment clinical studies and to elucidate mechanisms of resistance to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed advanced breast cancer (ABC), including locally advanced inoperable disease and stage IV disease.
2. Age > 18 years.
3. Performance status according to Eastern Cooperative Oncology Group (ECOG) ≤ 2.
4. ABC must be radiologically or clinically assessable, by means of at least one of the following techniques: clinical examination, computerized tomography (CT-scan), magnetic resonance imaging (MRI), bone scintigraphy or positron emission tomography (PET).
5. Patients must have a radiological evaluation done maximum 6 weeks prior to inclusion.
6. Signed informed consent according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

Untreated psychiatric disorders that will impair the patient's ability to comply with study treatment or protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic, inoperable breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years
  Prospective recording of treatment interventions and molecular characteristics in metastatic breast cancer patients until the date of Death.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University Hospital, Lund, Sweden